CLINICAL TRIAL: NCT05314452
Title: Timed Motor Function Test Using Video Based Observation and Online Based Observation Among Middle School Going Children: A Reliability and Validity Study
Brief Title: Reliability and Validity of 10 Meters Walk Test Among Children
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Professor, Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/2167
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: The Study Focuses to Find the Intrarater Reliability, Test-retest Reliability and Validity of 10 Meters Walk Test Among Middle School Going Children
Keywords: Child; Communication media; Health services; Reproducibility of results; Research design

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Timed Motor Function Tests (TMFTs) determined the walking abilities of an individual. During Covid-19 pandemic direct observation may not be feasible to record Timed motor function in children. Hence, the reliability and validity of video based observation and online based observation (VBO and OBO) methods to be explored. Middle school going children age group between 8 and 12 years was recruited for the study on the basis of convenience sampling. Sample size selected for each age group was according to sample size criteria of Interclass coefficient analysis. After anthropometrics, 10 meters walk test was recorded using three methods; VBO, OBO and direct observation for three times to estimate intrarater reliability and three days within a week to estimate test-retest reliability. The mean of three readings was used to find the estimated value. Direct observation method was used as a criterion measure method to report concurrent validity. After concurrent validity, Test-retest Reliability and Intrarater Reliability of VBO and OBO was reported. Reliability and validity of VBO and OBO with direct observation was reported by recording 10 meters walk test in children.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic middle school going children
2. Boys and girls in the age group between 8 and 12 years
3. Independent walking has achieved at age of 14 months
4. Able to understand and follow commands of examiner.

Exclusion Criteria:

1. Any Neurological disease
2. Any musculoskeletal disease in Lower Limb
3. Deformity in Lower Limb
4. Past history of surgery in Lower Limb in past 1 year
5. Any cardio-respiratory difficulties. -

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Middle school going children from tertiary school of Mullana-Ambala region
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
10 meters walk test (Direct observation method) | Immediate after taking anthropometric measurements
  10 meters walk test (TMFTs) determined the walking abilities of an individual using mobile phone stopwatch.
10 meters walk test (Video based observation method) | Immediate after measuring 10 meters walk test with direct observation method
  10 meters walk test using video camera of mobile phone
10 meters walk test (Online based observation method) | Immediate after measuring 10 meters walk test with Video based observation method
  10 meters walk test using online mobile based application- WhatsApp

CONTACTS AND LOCATIONS:
Overall Officials: Amit Kumar, (MPT), Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Asir John Samuel, PhD, Study Director — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Maharishi Markandeshwar International school, Ambāla, Ambala, India